### **Consent to Participate in Research**


**Title of Research Study:** Virtual Reality Job Interview Training: An Enhancement to

Supported Employment for Individuals with Severe Mental Illness; IRB# 202936

**Investigator:** Dr. Neil Jordan, Ph.D.

**Supported By:** This research is supported by National Institute of Mental Health.

#### **Key Information about this research study:**

The following is a short summary of this study to help you decide whether to be a part of this study. Information that is more detailed is listed later on in this form.

The purpose of this study is evaluate the process of implementing the Virtual Reality Job Interview Training (also known as "Molly") at Thresholds Inc. We are asking staff from the Employment Team to provide information to help us understand how implementing the Molly intervention into the Supported Employment Program went. Employment Specialists and Team Leaders will be asked to complete bi-weekly online surveys, participate in a focus group, and complete a short survey. Members of the Supported Employment Leadership Team will be asked to complete a short survey in the beginning of the study, and another survey in the middle of the study. We expect that you will be in this research study for the duration of the study, around 2 years.

#### Why am I being asked to take part in this research study?

We are asking you to take part in this research study because you are employed by Thresholds in the capacity as an Employment Coordinator or Employment Specialist within the Individual Placement and Support Program or you are in a leadership position within Thresholds such as a Manager, Director, or Officer.

### How many people will be in this study?

We expect approximately 20 staff, managers, directors, and leaders will be in this research study.

# What should I know about participating in a research study?

- Someone will explain the research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# What happens if I say, "Yes, I want to be in this research"?

- If you are part of the Supported Employment Leadership team:
  - Before delivery of the Molly intervention begins, we will ask you to complete a short, 12-item survey called the Implementation Leadership Scale. This survey should only take around 5 minutes and will help us understand your perspective on implementing evidence-based practice.
  - o After Molly has been delivered at Thresholds for 6 months, we will ask you to complete a 31item survey that will take approximately 20 minutes. These questions will ask about your views

#### **Consent to Participate in Research**


on the approach used by Thresholds to deliver the virtual reality training to participants, advantages of using the virtual reality training compared to typical services, and available resources that might help or hinder the implementation of the virtual reality training at Thesholds.

- If you are a Team Leader or Employment Specialist:
  - We will ask you to complete brief online survey (approximately 10 minutes to complete) every other week. This survey will ask about your time spent typical work activities and the implementation of the virtual reality training. This is known as the cost-capture survey. You will receive a link to this survey to your email every other Friday.
  - After virtual reality training has been delivered for several months at Thresholds, you may be asked to participate in a focus group that will last approximately 1 hour, to be conducted at Thresholds Inc. (4101 N. Ravenswood Ave, Chicago, IL 60613). The focus group will be facilitated by a Northwestern researcher. We will video-record the focus group to make sure that we do not miss or forget any of your feedback. We will transcribe the video record and then destroy the recording. To participate in the focus group, it is a requirement to be video-recorded.
  - At this time, we will also ask you to complete a 26-item Implementation Survey for Providers (<10 minutes) to gain your perspective on how integrating Molly into IPS is going.</li>

### Is there any way being in this study could be bad for me?

There are no known risks for this study as the surveys and questionnaires will be completed anonymously and the focus group will be facilitated by Northwestern University staff so your individual responses will not be available for any other staff, management, or leaders to view.

### What happens if I do not want to be in this research?

Participation in research is voluntary. You can decide to participate or not to participate.

## What happens if I say "Yes", but I change my mind later?

You can leave the research at any time and it will not be held against you. At any time in the study, you may decide to withdraw from the study. If you withdraw no more information will be collected from you and we will not contact you further. When you indicate you wish to withdraw the investigator will ask if the information or materials already collected from you can be used in the research analyses. If you do not want your study data to be used then you need to provide a formal, written request to the research team.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB, other representatives of this institution, as well as representatives of the National Institute of Mental Health and other University research centers and University contractors who are also working on the study.

A description of this clinical trial (NCT03049813) will be available at http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. This research is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH). This Certificate says that the researchers on this study cannot share or use information that may identify you in the event of a legal action or court proceeding. For example, if there is a court subpoena asking for your information from this study, the researcher cannot give your information to the court unless you consent to it. Your information is protected by this Certificate and cannot be shared with anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse); if you, yourself, have consented and agreed to share the information, including for your medical treatment; or if it is used for other scientific research (only when it is allowed by federal regulations protecting research subjects). The Certificate cannot be used to refuse a

**Document Template Revision Date: 4-6-2018** 

#### **Consent to Participate in Research**


request for information that is needed for auditing or program evaluation by NIH or for information that must be shared in order to meet the requirements of the Federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not stop you from voluntarily releasing information about yourself or your involvement in this research. If you want to share research information with an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. Unless you revoke your consent, it will expire at the close of the study. Data Sharing: De-identified data from this study may be shared with the research community at large to advance science and health. We will remove or code any personal information that could identify you before files are shared with other researchers to ensure that, by current scientific standards and known methods, no one will be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

#### Who can I talk to?

If you have questions, concerns, or complaints, you can talk to the person in charge of this study, Dr. Neil Jordan, at (312) 503-6137 or neil-jordan@northwestern.edu.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (312) 503-9338 or irb@northwestern.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.

Your signature documents your permission to take part in this research.

• You want to get information or provide input about this research.

### Signature for Adult 18 or older

| Signature of participant | Date | |
|------------------------------------------|------|---|
| Printed name of participant | | |
| Signature of person obtaining consent | Date | _ |
| Printed name of person obtaining consent | | |